CLINICAL TRIAL: NCT03617393
Title: A Prospective Study of Appropriate Technology of Standardized Diagnosis and Treatment for Diabetic Patients With Complication of Pulmonary Infection
Brief Title: Study on Appropriate Technology of Standardized Diagnosis and Treatment for Diabetic Patients With Pulmonary Infections
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, ZHOU Min, Chief Physician of Department of Respiratory Medicine, Ruijin Hospital
Other Study IDs: 2017YFC1309700
Record Dates: First submitted 2018-07-12; First posted 2018-08-06 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Diabetes Mellitus; Pulmonary Infection
Keywords: Early Warning Model; Clinical Pathway; Diabetes; Pulmonary Infection
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Pulmonary Infection with DM group: Patients with diabetes and pulmonary infection.
- Pulmonary Infection group: Patients with pulmonary infection while the fasting blood-glucose in the normal range.
- DM group: Patients without pulmonary infection while the fasting blood-glucose > 8 mmol/L.
- Control group: normal people: Patients without pulmonary infection while the fasting blood-glucose in the normal range.

SUMMARY:
Focusing on patients with diabetes complicated with pulmonary infection, the purpose of this study is: 1) to identify the epidemiology, etiologic spectrum and status of diagnosis and treatment; 2) to develop a symptom score scale , clarify the risk factors and create a precise warning model; 3) to develop a rapid detection of pathogen of lower respiratory infection, to establish clinical pathways of early diagnosis and treatment of diabetes complicated with pulmonary infections (including bacterial, tuberculosis and fungal infections) and then make an application in clinic.

DETAILED DESCRIPTION:
Investigators perform a observational study on 6000 patients with diabetes, among which 200 patients with pulmonary infection are included in a retrospective study and 100 patients go through metabolomics research. All patients receive clinical questionnaires, laboratory examinations and pulmonary function tests. Investigators study on pathogen distribution and infection ratio of patients above depending on follow-up survey. 1:1 nested case-control study is carried out involving 100 cases from pulmonary-infected group paired with 100 control cases matched for gender, age and fasting blood-glucose. The final purpose is to create a precise warning model in order to develop a rapid detection of pathogen of lower respiratory infection in diabetes patients. Now investigators wish to register this study to do a further research, in order to improve the early diagnosis of diabetes complicated with pulmonary infection and to reduce the mortality.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis by pathogen examination: positive
* Diagnosis through X-ray or CT: characteristic features of pulmonary infection
* Diagnosis through guideline of diabetes or history of diagnosed diabetes
* Age 40-70 years

Exclusion Criteria:

* Irregular follow-up and lost follow-up
* Withdraw from the study for any reason

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: diabetes patients complicated with pulmonary infection
Sampling Method: Non-Probability Sample
Enrollment: 6000 (Estimated)
Dates: Start 2017-07-10 (Actual); Primary Completion 2019-05-01 (Actual); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
Survival at 30 Days | 30 days from date of diagnosis of pulmonary infection until the date of death from any cause.
  Accuracy and sensitivity of novel survival prediction algorithm derived from differences between the predicted and actual 30-day-survival of patients from different groups.
Survival at 90 Days | 90 days from date of diagnosis of pulmonary infection until the date of death from any cause.
  Accuracy and sensitivity of novel survival prediction algorithm derived from differences between the predicted and actual 90-day-survival of patients from different groups.
Survival at 1 Year | 1 year from date of diagnosis of pulmonary infection until the date of death from any cause.
  Accuracy and sensitivity of novel survival prediction algorithm derived from differences between the predicted and actual 1-year-survival of patients from different groups.

SECONDARY OUTCOMES:
Hospitalization Time | Every 6 months from date of diagnosis of pulmonary infection until the date of death from any cause, assessed up to 3 years
  Differences in the time of hospital stay including ordinary sickroom and ICU of patients from different groups.
Sepsis | Every 6 months from date of diagnosis of pulmonary infection until the date of death from any cause, assessed up to 3 years
  Differences in the primary and secondary sepsis after therapy according to guideline from different groups.
CURB-65 Score | Every 6 months from date of diagnosis of pulmonary infection until the date of death from any cause, assessed up to 3 years
  Differences in confusion, urea, respiratory rate and age 65 scoring system from different groups.
Inflammatory Parameters | Day 0, day 3, day 10-14 and final result from date of diagnosis of pulmonary infection until the date of death or cure from any cause, assessed up to 1 years
  Differences in CRP, PCT, IL-6, IL-8, TNF-α from different groups.
Fungal Infection Examinations | Day 0, day 3, day 10-14 and final result from date of diagnosis of pulmonary infection until the date of death or cure from any cause, assessed up to 1 years
  Assessment of G test and GM test in order to clarify the diagnosis of fungal infection.
Cryptococcal Infection Examinations | Day 0, day 3, day 10-14 and final result from date of diagnosis of pulmonary infection until the date of death or cure from any cause, assessed up to 1 years
  Assessment latex agglutination test in order to clarify the cryptococcal infection.
Cell-mediated Immunoserologic Indexs | Day 0, day 3, day 10-14 and final result from date of diagnosis of pulmonary infection until the date of death or cure from any cause, assessed up to 1 years
  Differences of CD3, CD4 and CD8 in different groups in order to research on cell-mediated immunity of patients with or without diabetes and pulmonary infection.
Humoral Immunoserologic Indexes | Day 0, day 3, day 10-14 and final result from date of diagnosis of pulmonary infection until the date of death or cure from any cause, assessed up to 1 years
  Differences of IgG, IgA, IgE and IgM in different groups in order to research on cell-mediated immunity of patients with or without diabetes and pulmonary infection.

CONTACTS AND LOCATIONS:
Overall Officials: Jieming QU, Ph.D., M.D., Principal Investigator — China, Shanghai Ruijin Hospital Shanghai Jiao Tong University School of Medicine
Locations (1):
- Ruijin Hospital Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No